CLINICAL TRIAL: NCT06431659
Title: Swedish Palliative Care Guide (S-PCG) at Nursing Homes
Status: Enrolling by invitation | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00597-01, 2023-02274-01
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Age Problem; Old Age; Debility; Dementia
Keywords: Palliative care; Elderly; Nursing homes; Dementia
MeSH Terms: conditions — Frailty; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active group: The S-PCG is a person-centered decision support to identify, assess, document and meet palliative care needs and increase patients' quality of life and participation in their health-care decisions. The purpose of the S-PCG is to ensure the quality of care in continuous dialogue between health care staff, patient, and family, from the transition from curative to palliative care, to the patient dying, and the care afterwards. In the Care Guide, the patients' plans and wishes are documented, and based on this care be prioritized, planned, and coordinated. The S-PCG is adapted to be used throughout the health and medical care and in municipal care. The S-PCG consists of three parts that can be used separately, the intervention in this study includes S-PCG part 2 and 2D.
  In the active group the nursing homes will get our help to implement the S-PCG immediately, and data will be collected after the implementation.
- Control group: The S-PCG is a person-centered decision support to identify, assess, document and meet palliative care needs and increase patients' quality of life and participation in their health-care decisions. The purpose of the S-PCG is to ensure the quality of care in continuous dialogue between health care staff, patient, and family, from the transition from curative to palliative care, to the patient dying, and the care afterwards. In the Care Guide, the patients' plans and wishes are documented, and based on this care be prioritized, planned, and coordinated. The S-PCG is adapted to be used throughout the health and medical care and in municipal care. The S-PCG consists of three parts that can be used separately, the intervention in this study includes S-PCG part 2 and 2D.
  In the control group data will be collected before the implementation of S-PCG.

SUMMARY:
Palliative care aims to improve the quality of life for patients and families who are affected life-threatening, incurable disease. The care should be person-centred, but it is not entirely clear how this is best achieved. The Institute for Palliative Care, Lund, has developed the Swedish Palliative Care Guide (S-PCG) which support for a person-centred approach throughout the palliative care process.

The aim of this study is to improve palliative care for people living at nursing homes, including people with dementia and cognitive impairment, this will be achieved by providing support for health care staff working with this group of patients, investigating evidence for a palliative care the support tool, the Swedish Palliative Care Guide (S-PCG) part 2, and integrating the palliative care approach earlier in the disease trajectory, to improve the quality of care for this patient group. The research questions will be explored from the perspective of the patient, the family, and the staff.

DETAILED DESCRIPTION:
The study will include six-ten (based on number of patients in every cluster) nursing homes who are interested in implementing the S-PCG part 2. Among the included nursing homes half will be randomized to get help to implement the S-PCG immediately (active group), while the other half will get the same help somewhat later, and act as a control group until then (control group). The process of implementing S-PCG includes education and training in using the Care guide, this training is available physically as well as digitally. The implementation process, including education and training for staff, normally takes three months. To investigate the effect of the Care Guide among patients and families, a survey will be used among the patients' and their families at start of the study in the control group and after the end of the implementation period in the active group. The patients and family members who are willing to participate in the research will be asked to answer a one-page questionnaire about their experience of the care and about the future care. In patients that are not capable of an informed consent, we will only approach the families. All questions will be answered on a five-point Likert scale. The first part of the questionnaire (seven questions) are from the validated Swedish National Patient Survey and the other six questions are self-developed by the research group to explore the persons experience of planning of the care regarding to what extent they feel involved in the care, that the patient´s and relative´s wishes about future care are known to the health care professionals and that they can talk about end-of-life issues. Data from medical records will be collected regarding diagnoses, treatments, planning of treatment, communication, and restrictions of care (behandlingsbegränsningar).

Health care professionals (HCPs) will be asked to fill in a validated questionnaires about compassion fatigue among, the Compassion Fatigue Inventory (CFI) as HCPs are of high risk of fatigue. In the control group this will be performed at study start and in the control group after implementation of S-PCG. Moreover, HCPs in the active group are asked to participate in focus groups interviews regarding the implementation of the S-PCG and how it works in the clinical work.

Data collection: The cognitive function of patients will be evaluated by the HCPs together with the research staff and only those capable of writing an informed consent and answering the questionnaires will be included. Permission to ask a relative is done at inclusion. In those not able to consent, only relatives will be approached. Data will be collected from the questionnaire from patient and relatives. Questionnaires to patients will be performed on paper, together with a research person. The questionnaire will be read twice. Questionnaires to relatives will be given/sent by mail on paper, electronically or filled in by phone. Informed consent will be asked for at the same time, on paper, electronically or by phone (on tape). The questionnaires will be administered by the staff at the nursing homes and/or by staff at the Institute for Palliative Care, who will also digitalize the data. Data from questionnaires to HCPs will be given on paper or electronically as for relatives. Focus group interviews will be performed according to an interview guide at the nursing homes with 4-7 HCP participants, recorded and transcribed verbatim.

Analysis: The experiences of patients and relatives in nursing homes using the Care Guide (active group) will be compared with the experiences of families of patients in the control facilities included in the study, where the Care Guide is not yet implemented. The purpose of randomizing which nursing homes who implements the Care Guide first is to ensure that the difference that families may experience comes from the Care Guide itself, and not from the staff at a nursing home who choose to get involved and use a guide for good palliative care is better from the beginning, however adjustments of characteristics of the patients and setting might still be needed. The outcomes measured in this study is to which degree the patients and their families feel informed about the situation of the patient and their sense of security with the future care, after the Care Guide has been used.

ELIGIBILITY:
Inclusion Criteria:

- Living at one of the nursing homes that participates in the study and consents to the study or that next of kin consents (in case of excessively impaired cognition).

Exclusion criteria:

* That the person is dying or too ill to be asked about participation.
* That the person is not capable of giving their informed consent (e.g. due to their dementia) and missing relatives.

Ages: 65 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients living at nursing homes. Relatives to the included patients. Personal working at nursing homes
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2027-05-03 (Estimated); Study Completion 2028-05-03 (Estimated)

PRIMARY OUTCOMES:
To which degree the patients and their families feel informed about the situation of the patient. | Data will be collected through study completion, an average of 2 years, data will be collected only on time per patient.
  Measured by likert scale, 1-5. Higher number indicate higher experience of information.
To what degree the patients and their families feel secure about the future care that the patient will receive. | Data will be collected through study completion, an average of 2 years, data will be collected only on time per patient.
  Measured by likert scale, 1-5. Higher number indicate higher experience of security.

SECONDARY OUTCOMES:
Breakpoint conversation | Data will be collected through study completion, an average of 2 years, data will be collected only on time per patient.
  Presence of documented break point conversations in medical records.
Treatment limitations | Data will be collected through study completion, an average of 2 years, data will be collected only on time per patient.
  Presence of documented treatment limitations in medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Schelin, ass. prof., Principal Investigator — Region Skåne
Locations (1):
- Valgossens äldreboende, Stockholm, Region Stockholm, Sweden